CLINICAL TRIAL: NCT03602781
Title: Phase 3, Multicenter, Randomized, Double-blind, Placebo Controlled Withdrawal Study of Pulmonary Arterial Hypertension(PAH) Subjects With LTOT Use That Have Demonstrated Improved Exercise Tolerance With the Use of Inhaled Nitric Oxide (INO)
Brief Title: Study of PAH Subjects With LTOT Use That Have Demonstrated Improved Exercise Tolerance With the Use of Inhaled Nitric
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision not to proceed with Study
Sponsor: Bellerophon Pulse Technologies (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Organization: Bellerophon (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PULSE-PAH-007
Record Dates: First submitted 2018-07-06; First posted 2018-07-27 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2018-07

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; Inhaled Nitric Oxide; iNO; Long Term Oxygen Therapy; Oxygen therapy
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Nitrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Placebo 99.999% Nitrogen (Placebo Comparator): Randomized Withdrawal Treatment Period Week 1-8:
  Placebo at a dose setting of 75 mcg/kg IBW/hr for up to 24 hr/day
  Long Term Open Label Extension Period:
  iNO at a dose setting of 75 mcg/kg IBW/hr for up to 24 hr/day
  Interventions: Drug: Placebo; Drug: iNO
- Cohort 2: iNO 75 mcg/kg IBW/hr (Active Comparator): Randomized Withdrawal Treatment Period Week 1-8:
  iNO at a dose setting of 75 mcg/kg IBW/hr for up to 24 hr/day
  Long Term Open Label Extension Period:
  iNO at a dose setting of 75 mcg/kg IBW/hr for up to 24 hr/day
  Interventions: Drug: iNO

INTERVENTIONS:
Drug: Placebo — Placebo at a dose setting of 75 mcg/kg IBW/hr
  Other Names: Placebo 99.999% Nitrogen
  Arms: Cohort 1: Placebo 99.999% Nitrogen
Drug: iNO — iNO at a dose setting of 75 mcg/kg IBW/hr
  Other Names: Inhaled Nitric Oxide

SUMMARY:
Study of PAH Subjects with LTOT Use that have Demonstrated Improved Exercise Tolerance with the use of Inhaled Nitric Oxide

DETAILED DESCRIPTION:
Phase 3, Multicenter, Randomized, Double-blind, Placebo Controlled Withdrawal Study of Pulmonary Arterial Hypertension(PAH) Subjects with LTOT Use that have Demonstrated Improved Exercise Tolerance with the use of Inhaled Nitric Oxide (INO)

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form prior to the initiation of any study mandated procedures or assessments
2. Subjects must be enrolled in the PULSE PAH-004 clinical trial and must have been on LTOT and on open-label treatment with iNO 75 mcg/kg IBW/hr for at least 4 months
3. Subjects must have achieved ≥ 30 meter improvement in 6MWD after 4, 8 or 12 months of open-label treatment with iNO 75 mcg/kg IBW/hr as compared to either their PULSE PAH-004 Week 2 end of Run-in OR End of Study (EOS)in PULSE-PAH-004.
4. Subjects are willing and considered in the judgement of the Investigator able to use the INOpulse device continuously for up to 24 hours per day
5. Female subjects of childbearing potential must have a negative pregnancy test (serum or urine) at randomization. All female subjects must use an effective method of birth control to avoid pregnancy.

Exclusion Criteria:

1. Subjects with episodes of worsening of PAH in the last 30 days prior to PULSE PAH-007 Baseline/Randomization
2. Subjects that experience Pulmonary Rebound in PULSE-PAH-004
3. Change in dose or types of PAH specific therapies in the last 30 days prior to Baseline/Randomization
4. Subjects who require treatment with riociguat
5. Subjects who early discontinued drug/device usage due to withdrawal of consent or an adverse event requiring termination from treatment in PULSE PAH-004
6. Women who are pregnant
7. The concurrent use of the INOpulse device with a continuous airway pressure (CPAP), Bilevel Positive Airway Pressure (BiPAP, or any other positive pressure device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Time to clinical worsening during iNO withdrawal for up to 8 weeks | 8 weeks
  A clinical worsening event is defined as:
  1. Death (all-cause mortality)
  2. Atrial septostomy
  3. Hospitalization due to worsening of PAH
  4. Need to start additional specific PAH treatment
  5. Decrease of >15% in 6 Minute Walk Distance from randomization into the study
  6. Worsening of WHO Functional Class (e.g., from Class II to Class III or IV, OR Class III to Class IV)

SECONDARY OUTCOMES:
Difference in clinical worsening events that occur during iNO withdrawal for up to 8 weeks between those treated with iNO ≥ 10 months prior to the start of withdrawal of iNO vs. those treated < 10 months prior to initiation of withdrawal to iNO. | 8 weeks
  A clinical worsening event is defined as:
  1. Death (all-cause mortality)
  2. Atrial septostomy
  3. Hospitalization due to worsening of PAH
  4. Need to start additional specific PAH treatment
  5. Decrease of >15% in 6 Minute Walk Distance from randomization into the study
  6. Worsening of WHO Functional Class (e.g., from Class II to Class III or IV, OR Class III to Class IV)

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, MD, Study Director — Bellerophon Therapeutics
Locations (4):
- United States (2):
  - Bluhm Cardiovascular Institute, Clinical Trials Unit, Chicago, Illinois
  - Medical University of South Carolina, Charleston, South Carolina
- Canada (2):
  - Peter Lougheed Centre, Calgary, Alberta
  - Toronto General Hospital, University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No